CLINICAL TRIAL: NCT04754971
Title: Effectıveness Of Cognıtıve Behavıoral-Based Psychoeducatıon In College Students Wıth Smartphone Addıctıon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Ayse Tansu
Record Dates: First submitted 2021-02-12; First posted 2021-02-15 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Addictive Behavior
Keywords: Addiction, Smartphone; Cognitive Behavioral Therapy; Psychoeducation
MeSH Terms: conditions — Behavior, Addictive; Internet Addiction Disorder

STUDY DESIGN:
Intervention Model Description: Experimental design with pretest-posttest control group and follow-up measurements
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Table (Experimental)
  Interventions: Other: psycho-education program

INTERVENTIONS:
Other: psycho-education program — Psychoeducation Practice 1 day per week, 60-90 min. sessions will take 8 weeks. At the end of the training, the final test will be applied to the experimental and control group. 3rd and 6th month follow-up measurements are planned to be carried out intermittently at the end of the month.

SUMMARY:
This study aims to determine the effectiveness of the group psycho-education program which is prepared as "cognitive behavioural-based", on college students' smartphone dependency levels. The research will be carried out on students studying at a private foundation University in 2019-2020 academic year. In this study, pre-test-final Test control group and follow-up measured experimental pattern will be used to determine the effect of Psycho-education program on smartphone dependency levels of college students.

A Personal Information Form and Smartphone Dependency scale will be applied to students who agree to participate in the study. By analysing the data results obtained from the data collection tools and passing the determined limit value, 94 people will be randomly selected, including 47 experiments and 47 control groups, from those who scored high on the smartphone dependency scale through the SPSS program using the power analysis method. Students will be informed about cognitive behavioural based psychoeducation and will be asked if they wish to participate in the training. Psychoeducation Practice 1 day per week, 60-90 min. sessions will take 8 weeks. At the end of the training, the final test will be applied to the experimental and control group. 3rd and 6th month follow-up measurements are planned to be carried out intermittently at the end of the month.

In the literature, it is observed that the number of intervention studies is very small, and no clear conclusions have been reached. In addition, the treatment of smartphone addiction in Turkey with cognitive-behavioural approach-based group psychoeducation program has not been studied before. In our country, where smartphone addiction is increasing every day, the importance of intervention efforts in this area is clear. It is anticipated that the intervention study on addiction reduction will be supportive for researchers and will be beneficial for people who need support for smartphone addiction. In this respect, it is thought that it will be a guiding work for future clinical and academic studies.

ELIGIBILITY:
Inclusion Criteria:

Being over 18 years old Higher smartphone addiction scale score

Exclusion Criteria:

-

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-07-12 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Smartphone Addiction Scale-Short Form | 20 minutes
  mart Phone Addiction Scale Short Form: Smartphone Addiction Scale is a 6-point Likert-type scale consisting of 10 items developed by Kwon et al. (Kwon M, et al. 2013) to determine smartphone addiction in adolescents. Its Turkish validity and reliability were made by Noyan et al. Individuals read the items and how valid the items are for them, "1-I strongly disagree", "2-I do not agree", "3-I partially disagree", "4-I partially agree", "5- They make a decision by making a mark on a grading that includes "I agree", "6-Strongly agree" Scale scores range between 10-60. The higher the score obtained from the test, the higher the risk of addiction. The scale has a single factor and does not have subscales. The cut-off score is 31 for men and 33 for women (Kim S, Kim R. A, 2002). Those who score 31 points for male participants and 33 points for female participants are divided into two groups as 'smart phone addicts', and participants below these points are 'not smart phone addicts'.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Tanşu, Study Chair — PhD student
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)